CLINICAL TRIAL: NCT00004478
Title: Study of Droxidopa in Patients With Neurologic Hypotension
Brief Title: Droxidopa in Treating Patients With Neurogenic Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/14180; MTS-GCO-98-243-3-NE
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2008-09-18 (Estimated); Status verified 2008-09

CONDITIONS: Shy-Drager Syndrome; Orthostatic Hypotension
Keywords: Shy-Drager Syndrome; cardiovascular and respiratory diseases; neurologic and psychiatric disorders; orthostatic hypotension; rare disease
MeSH Terms: conditions — Shy-Drager Syndrome; Hypotension, Orthostatic; Respiratory Tract Diseases; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Droxidopa

INTERVENTIONS:
Drug: droxidopa

SUMMARY:
Please note that the continuation study can be found at http://clinicaltrials.gov/show/NCT00633880.

RATIONALE: Neurogenic hypotension is a fall in blood pressure that occurs when one moves from a lying down to a standing position or after eating a meal. It causes one to feel dizzy, light headed, and weak. Neurogenic hypotension is caused by a problem in the part of the nervous system that controls such functions as heart rate and blood pressure. Droxidopa, a drug that may increase blood pressure, may be an effective treatment for neurogenic hypotension.

PURPOSE: Clinical trial to study the effectiveness of droxidopa in treating patients who have neurogenic hypotension.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive escalating doses of droxidopa or placebo for 7-14 days. Patients undergo blood pressure measurements hourly in both supine and standing positions.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Orthostatic hypotension due to autonomic nervous system failure Fall in systolic blood pressure (supine to standing) of at least 20 mm Hg and diastolic blood pressure of at least 15 mm Hg AND Symptoms of hypotension such as dizziness, light-headedness, unsteadiness, dimming or blurred vision
* History of syncope or near-syncope

--Prior/Concurrent Therapy--

* Endocrine therapy: No concurrent adrenergics Concurrent fludrocortisone allowed
* Other: Concurrent indomethacin, support garments, and high salt diets allowed

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, MD, Study Chair — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Result] Kaufmann H, Saadia D, Voustianiouk A, Goldstein DS, Holmes C, Yahr MD, Nardin R, Freeman R. Norepinephrine precursor therapy in neurogenic orthostatic hypotension. Circulation. 2003 Aug 12;108(6):724-8. doi: 10.1161/01.CIR.0000083721.49847.D7. Epub 2003 Jul 28. PMID 12885750
- [Result] Goldstein DS, Holmes C, Kaufmann H, Freeman R. Clinical pharmacokinetics of the norepinephrine precursor L-threo-DOPS in primary chronic autonomic failure. Clin Auton Res. 2004 Dec;14(6):363-8. doi: 10.1007/s10286-004-0221-z. PMID 15666063